CLINICAL TRIAL: NCT03274388
Title: Influence of Individualized Nutritional Therapy Combined With Whole Body Electromyostimulation on Patients With Chronic Liver Disease
Brief Title: Whole Body Electromyostimulation and Nutritional Therapy for Patients With Chronic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMS Nutr chronLiver
Record Dates: First submitted 2017-06-01; First posted 2017-09-06 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: parallel group, controlled pilot study
Masking Description: Masking is not possible, since the "intervention" group receives exercise intervention in addition to protein-rich nutritional therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Intervention of protein-rich nutritional therapy and counseling
  Interventions: Procedure: nutritional therapy
- Intervention (Experimental): Intervention of protein-rich nutritional therapy and counseling combined with whole body electromyostimulation exercise training
  Interventions: Procedure: nutritional therapy; Procedure: WB-EMS combined with nutritional therapy

INTERVENTIONS:
Procedure: nutritional therapy — protein-rich nutritional therapy and counseling, during study period of 12 weeks
Procedure: WB-EMS combined with nutritional therapy — protein-rich nutritional therapy and counseling plus whole body electromyostimulation exercise training, twice a week for 20 min., during study period of 12 weeks
  Arms: Intervention

SUMMARY:
The purpose of this study is to explore the influence of an innovative combined therapy involving optimized protein-rich nutritional therapy and highly effective muscle training by personalized whole-body electromyostimulation (WB-EMS) exercise to improve muscle mass, strength and functionality, physical capacity, fatigue and quality of life of patients with chronic liver disease.

DETAILED DESCRIPTION:
In the course of chronic liver disease a systemic inflammatory reaction promotes mediators leading to a loss of appetite, as well as to metabolic and hormonal changes. Consequences hereof are a decreased food uptake, a deteriorated nutrient utilization and a loss of muscles, with or without fat loss leading to cachexia. Especially muscle loss has a relevant influence on morbidity and mortality of chronic liver patients. The loss of muscle is probably due to a deteriorated protein synthesis with concurrent anabolic resistance. These pathologic processes increase the protein requirements of chronic liver patients dramatically.

The purpose of this study is to establish an innovative combined therapy involving optimized nutritional therapy and highly effective muscle training by personalized whole-body electromyostimulation (WB-EMS) exercise to improve the quality of life (QLQ) of patients with serious chronic disease. An improvement of QLQ results from an increase in muscle mass and strength, thereby increasing physical activity, physical capability as well as tolerance to and applicability of therapy. In the course of a 3-months intervention study the efficacy of a combined German-guidelines-recommended protein-rich nutritional therapy with an innovative exercise therapy will be documented for patients with chronic liver disease. An effective stopping of the progress of muscle wasting or even increase of muscle mass, strength and function in the patients of the trial would benefit each patient and his family individually, since it could mean a considerable improvement in his QLQ and tolerability of therapeutical treatment.

ELIGIBILITY:
Inclusion Criteria:

• Patients with chronic liver disease in curative or palliative treatment

Exclusion Criteria:

* Healthy persons or patients under age
* Pregnancy, Lactation,
* Psychological disorders, epilepsy, sever neurological disorders
* Participation in other exercise- or nutrition studies within the last 6 months
* acute cardiovascular disease
* Rheuma
* Intake of anabolic drugs,
* Skin injuries in the area of electrode placements
* Electronic implants (defibrillator, pacemaker)
* Persons in mental hospitals by order of authorities or jurisdiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Muscle mass of chronic liver patients | 3 months
  Increase or stabilization of muscle mass of chronic liver patients due to combinatorial therapy of protein-rich nutrition and WB-EMS. Muscle mass will be measured by Bioelectrical Impedance Analysis.
Muscle strength of chronic liver patients. | 3 months
  Increase or stabilization of muscle strength of chronic liver patients due to combinatorial therapy of protein-rich nutrition and WB-EMS. Muscle strength will be measured by hand grip strength measurements.

SECONDARY OUTCOMES:
Quality of life score as assessed by EORTC-QLQ-C30 | 3 months
  Increase or stabilization of quality of life score of chronic liver patients due to combinatorial therapy of protein-rich nutrition and WB-EMS.
Pain score as assessed by visual analogue score | 3 months
  Increase or stabilization of pain score of chronic liver patients due to combinatorial therapy of protein-rich nutrition and WB-EMS.
Fatigue score as assessed by FACIT-Fatigue-Score analysis | 3 months
  Increase or stabilization of fatigue score of chronic liver patients due to combinatorial therapy of protein-rich nutrition and WB-EMS.
Degree of toxicity of chemotherapy regarding gastrointestinal complaints as assessed by Common Toxicity Criteria (CTC) | 3 months
  Decrease of common toxicity criteria regarding gastrointestinal complaints of chronic liver patients due to combinatorial therapy of protein-rich nutrition and WB-EMS.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdaguel Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

REFERENCES:
- [Background] Plauth M, Schuetz, T, Pirlich, M, Canbay, A, DGEM Steering Committee. S3-Leitlinie der DGEM in zusammenarbeit mit der GESKES, der AKE und der DGVS_ Klinische Ernährung in der Gastroenterologie (Teil1) - Leber. Aktuelle Ernaehrungsmedizin 39: e1-e42, 2014